CLINICAL TRIAL: NCT01468610
Title: Neurocognition and Work Productivity in Major Depressive Disorder
Brief Title: Neurocognition and Work Productivity in Major Depressive Disorder (MDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11-02646; WS2087153 (Other Grant/Funding Number: Pfizer Canada Inc.)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Major Depressive Disorder
Keywords: depression; cognition; occupational functioning; productivity; neuropsychology; desvenlafaxine; antidepressants
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Workers with MDD (Active Comparator)
  Interventions: Drug: desvenlafaxine

INTERVENTIONS:
Drug: desvenlafaxine — 50-100 mg daily for 8 weeks
  Other Names: Pristiq

SUMMARY:
This study will investigate the relationships between subjective cognitive complaints, neurocognitive deficits, and work productivity in participants with Major Depressive Disorder (MDD), before and after 8 weeks of treatment with an antidepressant medication. Our hypothesis is that, in working participants with MDD of at least moderate severity, neurocognitive deficits will predict poorer work functioning and productivity.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Major Depressive Disorder as per DSM-IV-TR
2. Current employment of at least 15 hours per week
3. Baseline score of 23 or greater on the Montgomery-Asberg Depression Rating Scale, indicating at least moderately severe depression
4. Baseline score of 6 or greater on the British Columbia Cognitive Complaints Inventory, indicating at least moderate subjective cognitive complaints
5. Competency to give informed consent

Exclusion Criteria:

1. Current receipt of short-term or long-term disability benefits from employer
2. Serious suicidal risks as judged by the investigators
3. Other DSM-IV-TR diagnoses:

   1. organic mental disorders
   2. active substance abuse/dependence, including alcohol
   3. schizophrenia, paranoid or delusional disorders, or other psychotic disorders
   4. (as primary diagnosis:) panic disorder, generalized anxiety disorder, obsessive-compulsive disorder, or post-traumatic stress disorder
   5. bipolar disorder
   6. bulimia nervosa or anorexia nervosa
4. Serious illness that is not stabilized, including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic, or hematologic disease
5. Regular/current use of other psychotropic drugs and/or herbaceuticals
6. Use of fluoxetine within 5 weeks of Visit 1, monoamine oxidase inhibitors within 14 days of Visit 1, and other antidepressants within 7 days of Visit 1 (all to ensure adequate drug washouts prior to neurocognitive assessment)
7. Previous treatment with desvenlafaxine
8. Treatment-resistance in the current episode, as defined by failure (i.e., lack of clinically significant response) of 2 or more antidepressants given at therapeutic doses for at least 6 weeks
9. Any history of treatment with electroconvulsive therapy
10. Initiation of formal psychotherapy (e.g., cognitive-behavioural therapy or interpersonal psychotherapy) with 2 months of Visit 1, or plans to start such psychotherapy during this study
11. Current use of any other form of treatment for depression

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
cognitive functioning as determined by neuropsychological testing | change from baseline to 8 weeks
  Neuropsychological testing in 5 domains (memory, psychomotor speed, reaction time, cognitive flexibility, and complex attention) is conducted using computerized measures, both at baseline and after 8 weeks of standard medical care involving antidepressant medication (flexibly-dosed desvenlafaxine)

SECONDARY OUTCOMES:
work productivity as determined by rating scales | change from baseline to 8 weeks
  Work functioning (attendance and productivity) is assessed using subjective and objective measures, both at baseline and after 8 weeks of standard medical care involving antidepressant medication (flexibly-dosed desvenlafaxine)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond W Lam, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Department of Psychiatry, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Alonso-Prieto E, Rubino C, Lucey M, Evans VC, Tam EM, Woo C, Iverson GL, Chakrabarty T, Yatham LN, Lam RW. Relationship between work functioning and self-reported cognitive complaints in patients with major depressive disorder treated with desvenlafaxine. Psychiatry Res. 2019 Feb;272:144-148. doi: 10.1016/j.psychres.2018.12.062. Epub 2018 Dec 10. PMID 30583256
- [Derived] Sarfati D, Evans VC, Tam EM, Woo C, Iverson GL, Yatham LN, Lam RW. The impact of fatigue and energy on work functioning and impairment in patients with major depressive disorder treated with desvenlafaxine. Int Clin Psychopharmacol. 2017 Nov;32(6):343-349. doi: 10.1097/YIC.0000000000000192. PMID 28763344
- [Derived] Lam RW, Iverson GL, Evans VC, Yatham LN, Stewart K, Tam EM, Axler A, Woo C. The effects of desvenlafaxine on neurocognitive and work functioning in employed outpatients with major depressive disorder. J Affect Disord. 2016 Oct;203:55-61. doi: 10.1016/j.jad.2016.05.074. Epub 2016 May 31. PMID 27280963
- See also: University of British Columbia — http://www.ubc.ca